CLINICAL TRIAL: NCT07283835
Title: A Single-arm, Open-label, Multicenter Phase II Clinical Study to Evaluate the Efficacy and Safety of Cretostimogene Grenadenorepvec in Patients With BCG-unresponsive High-risk Non-Muscle Invasive Bladder Cancer
Brief Title: Study of Cretostimogene Given in Patients With Non-Muscle Invasive Bladder Cancer ,Unresponsive to Bacillus-Calmette-Guerin
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lepu Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG0070-II-CIS-01
Record Dates: First submitted 2025-12-06; First posted 2025-12-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non Muscle Invasive Bladder Cancer; High-grade Ta/ T1 Papillary Disease Bladder Cancer
Keywords: high-grade Ta papillary disease; high-grade T1 papillary disease; carcinoma in situ; Bacillus-Calmette-Guerin unresponsive
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma in Situ | interventions — dodecyl maltoside

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cretostimogene (Experimental): Patients with CIS with or without HG Ta/T1 papillary disease. Cretostimogene will be administered intravesically following a series of bladder washes with 5% DDM and normal saline. Cretostimogene will be administered weekly for specific schedule per protocol.
  Interventions: Biological: Cretostimogene Grenadenorepvec; Other: n-dodecyl-B-D-maltoside

INTERVENTIONS:
Biological: Cretostimogene Grenadenorepvec — Engineered Oncolytic Adenovirus
  Other Names: CG0070
Other: n-dodecyl-B-D-maltoside — Transduction-enhancing agent
  Other Names: DDM

SUMMARY:
This study aims to evaluate the efficacy and safety of Cretostimogene in patients with BCG-unresponsive high-risk non-muscle invasive bladder cancer (NMIBC) with carcinoma in situ (CIS), with or without Ta/T1 papillary tumors.

DETAILED DESCRIPTION:
An open-label trial designed to evaluate Cretostimogene + DDM in patients with NMIBC who have failed prior BCG therapy. Single treatment arm that enrolled patients with carcinoma in situ with or without concomitant high-grade Ta or T1 papillary disease.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the patient must:

1. Be ≥18 years of age on day of signing informed consent.

   - Patients must have pathologically confirmed BCG-unresponsive non-muscle-invasive bladder cancer (NMIBC) with carcinoma in situ (CIS), with or without concomitant Ta/T1 papillary disease.
2. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
3. Have all Ta and/or T1 disease resected and all CIS resected or fulgurated, as feasible, prior to study treatment.
4. Demonstrate adequate organ function.
5. Patients must be willing to comply with study mandated cystoscopies, urine cytology, urograms, biopsies, and other procedures (including TURBT or other resection for all Ta/T1 disease) for the duration of the study. Patients who withdraw consent for these procedures will be withdrawn from the trial.
6. Ineligible to receive radical cystectomy or refusal of radical cystectomy according to Investigator assessment.

Exclusion Criteria:

1. Has current or past history of muscle invasive (T2 or higher stage) or locally advanced (T3/T4, any N) or metastatic bladder cancer.
2. History of urothelial carcinoma in the upper genitourinary tract (kidney, renal collecting system, ureter) or in the prostatic urethra, including urethral CIS, within 24 months prior to enrollment.
3. Has received systemic anti-cancer therapy, including investigational agents.
4. Has had prior systemic treatment (with the exception of checkpoint inhibitor therapy), radiation therapy, or surgery for bladder cancer other than TURBT or bladder biopsies.
5. Has any of the following within the 6 months prior to starting study treatment: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, pulmonary embolus, uncontrolled hypertension, or uncontrolled congestive heart failure.
6. Cannot tolerate study-related biopsies, IVE administration, or 1-hour bladder hold of Cretostimogene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate at any time in BCG-unresponsive high-risk NMIBC with or without Ta/T1 papillary tumors including CIS | 36 months

SECONDARY OUTCOMES:
Duration of response (DOR) | 36 months
  Time from first documented objective response to disease progression or death from any cause.
Assess high-grade reoccurrence free survival (RFS) | 36 months
  Time from first treatment to first recurrence of high-grade disease or death from any cause.
Assess progression free survival (PFS) | 36 months
  Time from first treatment to tumor progression or death from any cause.
Complete response rate at 12, 24, and 36 months | Assessed at 12, 24, and 36 months
  Proportion of patients achieving complete response at 12, 24, and 36 months.
Overall survival rate at 36 months | 36 months
  Proportion of patients alive at 36 months.
Safety: incidence and severity of adverse events (AE) and serious adverse events (SAE) | 36 months
  Safety is evaluated based on NCI-CTCAE v5.0 criteria. This includes incidence and severity of all adverse events (AE), serious adverse events (SAE), and abnormal laboratory values.

CONTACTS AND LOCATIONS:
Overall Officials: Dinɡwei Ye, M.D., Principal Investigator — Fudan University
Locations (15):
- China (15):
  - Peking University First Hospital (First Clinical Medical School of Peking University), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No